CLINICAL TRIAL: NCT07231328
Title: Post-Transplant Application of TruGraf and TRAC Molecular Panel in Renal Transplant Recipients
Brief Title: PIONEER Trial (Post-Transplant Application of TruGraf and TRAC Molecular Panel in Renal Transplant Recipients)
Acronym: PIONEER
Status: Not yet recruiting | Type: Observational
Sponsor: Transplant Genomics, Inc. (Industry)
Collaborators: Medical University of South Carolina (Other); Northwestern University (Other); The Cleveland Clinic (Other); University of Washington (Other); University of California, Los Angeles (Other); University of Nebraska (Other); Duke University (Other); University of Utah (Other); Georgetown University (Other); Virginia Commonwealth University (Other); The Methodist Hospital Research Institute (Other); Keck School of Medicine USC (Unknown); Weill Medical College of Cornell University (Other); Erie County Medical Center (Other); East Carolina University (Other); AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: TGRP20_PIONEER
Record Dates: First submitted 2025-09-22; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Immunosuppression Management; Biomarkers / Blood; Subclinical Rejection; Biopsy; Kidney Transplant Rejection
Keywords: TRAC-ID ASSAY; Kidney Transplant rejection; TruGraf, TRAC/TRAC ID biomarker panel; TruGraf; TRAC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Natural History Subgroup
  Interventions: Diagnostic Test: There is no required Intervention for this Protocol. Based on Results for TruGraf/TRAC/TRAC ID Investigators may use the results in managing subjects Immunosuppression or rule out rejection.
- • Real-World Use Subgroup
  Interventions: Diagnostic Test: There is no required Intervention for this Protocol. Based on Results for TruGraf/TRAC/TRAC ID Investigators may use the results in managing subjects Immunosuppression or rule out rejection.

INTERVENTIONS:
Diagnostic Test: There is no required Intervention for this Protocol. Based on Results for TruGraf/TRAC/TRAC ID Investigators may use the results in managing subjects Immunosuppression or rule out rejection. — Investigators will prospectively record whether each results led to a change in clinical management. Participating sites will be encouraged to follow their usual practice, supplemented where appropriate by the suggested TruGraf and TRAC™ TRAC ID algorithms

SUMMARY:
This is an observational, prospective, multi-center trial designed to evaluate clinical outcomes in kidney transplant recipients undergoing TruGraf and TRAC monitoring.

Approximately 15 U.S. sites

DETAILED DESCRIPTION:
All subjects who meet the inclusion criteria and none of the exclusion criteria will be eligible to participate. As the study is non-interventional, no protocol-mandated treatment or management plan will be imposed. In the absence of a universally ac-cepted paradigm for post-transplant monitoring with molecular diagnostics, participat-ing sites will be encouraged to follow their usual practice, supplemented where ap-propriate by the suggested TruGraf and TRAC™ algorithms.

To evaluate both the prognostic performance and the clinical utility of these bi-omarkers, a hybrid analytic framework will be used. Biomarker results will be made available to clinicians in real time, and investigators will prospectively record whether each result led to a change in clinical management. Natural History Subgroup: Test-ing events in which both TruGraf® and TRAC results are double-negative and no change in management occurred. Analyses will be anchored at the test-event level to avoid immortal time bias. This subgroup will be used to evaluate the safety and true negative predictive value (NPV) of a double-negative result, including the incidence of biopsy-proven acute rejection (BPAR) within 30 days.

• Real-World Use Subgroup: Testing events in which biomarker results prompt-ed a change in clinical management (e.g., change in immunosuppression, for-cause biopsy, or enhanced monitoring). By definition, any action following a test result places the event in this subgroup, irrespective of whether the bi-omarker result was double-negative or abnormal. Because clinical actions can alter subsequent risk trajectories, analyses in this subgroup will account for treatment-confounder feedback using causal modeling strategies (e.g., marginal structural models, target trial emulation).

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the key components of the study as described in the written informed consent document and willing and able to provide written informed consent.
* At least 18 years of age at the time of screening.
* Enrollment begins 30 days prior to transplant till day 29 post-transplantation.
* Recipient of a kidney transplant (either primary or repeat), from either deceased or living donor.
* Receiving any immunosuppressive regimen.
* Able and willing to comply with all study procedures, as assessed by the Investigator.
* Selected by the treating provider to undergo TruGraf and TRAC™ testing as part of routine post-transplant care

Exclusion Criteria:

History of previous non-kidney solid organ, vascular composite allograft, pancreatic islet, stem cell, or bone marrow transplant.

* History of dual or en-bloc kidney transplants.
* Recipient or donor with positive test for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis B virus (HBV) nucleic acid testing (NAT), hepatitis C virus (HCV) antibody, HCV NAT, human immunodeficiency virus (HIV), or HIV NAT.
* Patients known to be pregnant or with plans to become pregnant over the 24 months after enrollment.
* History or presence of coagulopathy, thrombophilia, unexplained bleeding or clotting disorders, or use of or documented plans for use of systemic anticoagulants at the time of screening, with the exception of uremic coagulopathy or prophylactic heparin preparations.
* History or presence, upon clinical evaluation, of any illness or condition that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population- Post kidney transplant subjects 18 and older at leas 30 days post surgery will undergo TruGraf, TRAC and TRAC-ID biomarker testing at Mo 1,4,7,10,12,16,20 and 24.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate post-transplant clinical outcomes in recipients of kidney transplants who are undergoing TruGraf and TRAC™ monitoring | 24 Months post transplant
  The primary endpoint is a composite at 24-months post-transplant, defined as the occurrence of any of the following events:
  • Biopsy-proven acute rejection (BPAR) on any for-cause biopsy between Month 1 to Month 24 (local read).
  OR
  • De novo Class I or Class II DSA detected at Month 12 or Month 24 (centrally read).
  OR • Decline in eGFR ≥20% from Month 3 to Month 24, calculated using the CKD-EPI creatinine-based equation.
  OR
  • Three or more abnormal TruGraf and TRAC results between Months 1 and 24

SECONDARY OUTCOMES:
To evaluate the overall safety of TruGraf and TRAC monitoring in post-transplant recipients of kidney transplants. | Month 3 to Mo 24 post transplant
  Actions taken based on tests results TruGraf, TRAC/TRAC-ID
To asses the safety of a double negative TruGraf/TRAC result | Month 3 to Mo 24 post transplant
  Quantifying the incidence of biopsy -proven acute rejection (BPAR) withing 30 days among patients for whom no change in clinical management was undertaken
To explore the impact of biomarker -informed clinical decision-making on outcomes such as BPAR, estimated glomerular filtration rate (eGFR) trajectory, and immunosuppressive adjustments | Month 3 to Mo 24 post transplant
  Quantifying the incidence of biopsy -proven acute rejection (BPAR) withing 30 days among patients for whom no change in clinical management was undertaken

OTHER OUTCOMES:
Exploratory objective: Evaluate the utility of serial TRAC-ID assays to monitor viral or systemic infections and guide safe adjustments of immunosuppression | Mont 3- Mo 24
  TRAC-ID results will be available for Investigators

CONTACTS AND LOCATIONS:
Overall Officials: Isioma Agboli, MD, Study Director — Transplant Genomics

IPD SHARING:
Plan to Share IPD: No
Results and Statistical analysis will be shared with PI's and Internal steering committee for Journal publications. It will become available upon publications

REFERENCES:
- [Background] Clinical Utility of Peripheral Blood Gene Expression Profiling of Kidney Transplant Recipients to Assess the Need for Surveillance Biopsies in Subjects with Stable Renal Function January 2017 Journal of Transplantation Technologies & Research 07(03) DOI: 10.4172/2161-0991.1000177 Martin Roy First Thomas C Whisenant John Friedewald Show all 10 authors Michael M Abecassis Citations 6 Reads 239
- [Background] Analytical and Clinical Validation of a Molecular Diagnostic Signature in Kidney Transplant Recipients January 2017 Journal of Transplantation Technologies & Research 07(03) DOI: 10.4172/2161-0991.1000176
- [Background] Lo DJ, Kaplan B, Kirk AD. Biomarkers for kidney transplant rejection. Nat Rev Nephrol. 2014 Apr;10(4):215-25. doi: 10.1038/nrneph.2013.281. Epub 2014 Jan 21. PMID 24445740
- [Background] Bouamar R, Shuker N, Hesselink DA, Weimar W, Ekberg H, Kaplan B, Bernasconi C, van Gelder T. Tacrolimus predose concentrations do not predict the risk of acute rejection after renal transplantation: a pooled analysis from three randomized-controlled clinical trials(dagger). Am J Transplant. 2013 May;13(5):1253-61. doi: 10.1111/ajt.12191. Epub 2013 Mar 8. PMID 23480233
- [Background] Loupy A, Vernerey D, Tinel C, Aubert O, Duong van Huyen JP, Rabant M, Verine J, Nochy D, Empana JP, Martinez F, Glotz D, Jouven X, Legendre C, Lefaucheur C. Subclinical Rejection Phenotypes at 1 Year Post-Transplant and Outcome of Kidney Allografts. J Am Soc Nephrol. 2015 Jul;26(7):1721-31. doi: 10.1681/ASN.2014040399. Epub 2015 Jan 2. PMID 25556173
- [Background] Heilman RL, Devarapalli Y, Chakkera HA, Mekeel KL, Moss AA, Mulligan DC, Mazur MJ, Hamawi K, Williams JW, Reddy KS. Impact of subclinical inflammation on the development of interstitial fibrosis and tubular atrophy in kidney transplant recipients. Am J Transplant. 2010 Mar;10(3):563-70. doi: 10.1111/j.1600-6143.2009.02966.x. Epub 2010 Feb 1. PMID 20121731
- [Background] Mehta RB, Tandukar S, Jorgensen D, Randhawa P, Sood P, Puttarajappa C, Zeevi A, Tevar AD, Hariharan S. Early subclinical tubulitis and interstitial inflammation in kidney transplantation have adverse clinical implications. Kidney Int. 2020 Aug;98(2):436-447. doi: 10.1016/j.kint.2020.03.028. Epub 2020 Apr 25. PMID 32624181
- [Background] Mehta R, Bhusal S, Randhawa P, Sood P, Cherukuri A, Wu C, Puttarajappa C, Hoffman W, Shah N, Mangiola M, Zeevi A, Tevar AD, Hariharan S. Short-term adverse effects of early subclinical allograft inflammation in kidney transplant recipients with a rapid steroid withdrawal protocol. Am J Transplant. 2018 Jul;18(7):1710-1717. doi: 10.1111/ajt.14627. Epub 2018 Jan 17. PMID 29247472
- [Background] Arias M, Seron D, Herrero I, Rush DN, Wiebe C, Nickerson PW, Ussetti P, Rodrigo E, de Cos MA. Subclinical Antibody-Mediated Rejection. Transplantation. 2017 Jun;101(6S Suppl 1):S1-S18. doi: 10.1097/TP.0000000000001735. No abstract available. PMID 28538291
- [Background] Seifert ME, Yanik MV, Feig DI, Hauptfeld-Dolejsek V, Mroczek-Musulman EC, Kelly DR, Rosenblum F, Mannon RB. Subclinical inflammation phenotypes and long-term outcomes after pediatric kidney transplantation. Am J Transplant. 2018 Sep;18(9):2189-2199. doi: 10.1111/ajt.14933. Epub 2018 Jun 27. PMID 29766640
- [Background] Nankivell BJ, Agrawal N, Sharma A, Taverniti A, P'Ng CH, Shingde M, Wong G, Chapman JR. The clinical and pathological significance of borderline T cell-mediated rejection. Am J Transplant. 2019 May;19(5):1452-1463. doi: 10.1111/ajt.15197. Epub 2019 Jan 22. PMID 30501008
- [Background] Meier-Kriesche HU, Schold JD, Srinivas TR, Kaplan B. Lack of improvement in renal allograft survival despite a marked decrease in acute rejection rates over the most recent era. Am J Transplant. 2004 Mar;4(3):378-83. doi: 10.1111/j.1600-6143.2004.00332.x. PMID 14961990
- [Background] Saran R, Robinson B, Abbott KC, Agodoa LY, Albertus P, Ayanian J, Balkrishnan R, Bragg-Gresham J, Cao J, Chen JL, Cope E, Dharmarajan S, Dietrich X, Eckard A, Eggers PW, Gaber C, Gillen D, Gipson D, Gu H, Hailpern SM, Hall YN, Han Y, He K, Hebert H, Helmuth M, Herman W, Heung M, Hutton D, Jacobsen SJ, Ji N, Jin Y, Kalantar-Zadeh K, Kapke A, Katz R, Kovesdy CP, Kurtz V, Lavalee D, Li Y, Lu Y, McCullough K, Molnar MZ, Montez-Rath M, Morgenstern H, Mu Q, Mukhopadhyay P, Nallamothu B, Nguyen DV, Norris KC, O'Hare AM, Obi Y, Pearson J, Pisoni R, Plattner B, Port FK, Potukuchi P, Rao P, Ratkowiak K, Ravel V, Ray D, Rhee CM, Schaubel DE, Selewski DT, Shaw S, Shi J, Shieu M, Sim JJ, Song P, Soohoo M, Steffick D, Streja E, Tamura MK, Tentori F, Tilea A, Tong L, Turf M, Wang D, Wang M, Woodside K, Wyncott A, Xin X, Zang W, Zepel L, Zhang S, Zho H, Hirth RA, Shahinian V. US Renal Data System 2016 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2017 Mar;69(3 Suppl 1):A7-A8. doi: 10.1053/j.ajkd.2016.12.004. No abstract available. PMID 28236831
- [Background] Tonelli M, Wiebe N, Knoll G, Bello A, Browne S, Jadhav D, Klarenbach S, Gill J. Systematic review: kidney transplantation compared with dialysis in clinically relevant outcomes. Am J Transplant. 2011 Oct;11(10):2093-109. doi: 10.1111/j.1600-6143.2011.03686.x. Epub 2011 Aug 30. PMID 21883901
- [Background] Peddi VR, Patel PS, Schieve C, Rose S, First MR. Serial Peripheral Blood Gene Expression Profiling to Assess Immune Quiescence in Kidney Transplant Recipients with Stable Renal Function. Ann Transplant. 2020 Apr 28;25:e920839. doi: 10.12659/AOT.920839. PMID 32341330
- [Background] Loupy A, Haas M, Roufosse C, Naesens M, Adam B, Afrouzian M, Akalin E, Alachkar N, Bagnasco S, Becker JU, Cornell LD, Clahsen-van Groningen MC, Demetris AJ, Dragun D, Duong van Huyen JP, Farris AB, Fogo AB, Gibson IW, Glotz D, Gueguen J, Kikic Z, Kozakowski N, Kraus E, Lefaucheur C, Liapis H, Mannon RB, Montgomery RA, Nankivell BJ, Nickeleit V, Nickerson P, Rabant M, Racusen L, Randhawa P, Robin B, Rosales IA, Sapir-Pichhadze R, Schinstock CA, Seron D, Singh HK, Smith RN, Stegall MD, Zeevi A, Solez K, Colvin RB, Mengel M. The Banff 2019 Kidney Meeting Report (I): Updates on and clarification of criteria for T cell- and antibody-mediated rejection. Am J Transplant. 2020 Sep;20(9):2318-2331. doi: 10.1111/ajt.15898. Epub 2020 May 28. PMID 32463180
- [Background] Lee H, Colby C. Heat of polymerization of nine mono-, di-, and trimethacrylate esters tested neat and with low levels of peroxide by dynamic differential scanning calorimetry. Dent Mater. 1986 Aug;2(4):175-8. doi: 10.1016/s0109-5641(86)80031-8. No abstract available. PMID 3462064
- [Background] Arms MA, Fleming J, Sangani DB, Nadig SN, McGillicuddy JW, Taber DJ. Incidence and impact of adverse drug events contributing to hospital readmissions in kidney transplant recipients. Surgery. 2018 Feb;163(2):430-435. doi: 10.1016/j.surg.2017.09.027. Epub 2017 Nov 22. PMID 29174434
- [Background] Sinha R, Zhu Z, Park S, Rebello C, Kinsella B, Friedewald J, Kleiboeker S. Combined Metagenomic Viral Detection and Donor-Derived Cell-Free DNA Quantification in Plasma From Kidney Transplant Recipients. Transplant Proc. 2024 Jul-Aug;56(6):1522-1530. doi: 10.1016/j.transproceed.2024.06.003. Epub 2024 Jul 6. PMID 38972761
- [Background] Park S, Guo K, Heilman RL, Poggio ED, Taber DJ, Marsh CL, Kurian SM, Kleiboeker S, Weems J, Holman J, Zhao L, Sinha R, Brietigam S, Rebello C, Abecassis MM, Friedewald JJ. Combining Blood Gene Expression and Cellfree DNA to Diagnose Subclinical Rejection in Kidney Transplant Recipients. Clin J Am Soc Nephrol. 2021 Oct;16(10):1539-1551. doi: 10.2215/CJN.05530421. PMID 34620649
- [Background] Zhang W, Yi Z, Keung KL, Shang H, Wei C, Cravedi P, Sun Z, Xi C, Woytovich C, Farouk S, Huang W, Banu K, Gallon L, Magee CN, Najafian N, Samaniego M, Djamali A, Alexander SI, Rosales IA, Smith RN, Xiang J, Lerut E, Kuypers D, Naesens M, O'Connell PJ, Colvin R, Menon MC, Murphy B. A Peripheral Blood Gene Expression Signature to Diagnose Subclinical Acute Rejection. J Am Soc Nephrol. 2019 Aug;30(8):1481-1494. doi: 10.1681/ASN.2018111098. Epub 2019 Jul 5. PMID 31278196
- [Background] Friedewald JJ, Kurian SM, Heilman RL, Whisenant TC, Poggio ED, Marsh C, Baliga P, Odim J, Brown MM, Ikle DN, Armstrong BD, Charette JI, Brietigam SS, Sustento-Reodica N, Zhao L, Kandpal M, Salomon DR, Abecassis MM; Clinical Trials in Organ Transplantation 08 (CTOT-08). Development and clinical validity of a novel blood-based molecular biomarker for subclinical acute rejection following kidney transplant. Am J Transplant. 2019 Jan;19(1):98-109. doi: 10.1111/ajt.15011. Epub 2018 Aug 31. PMID 29985559
- See also: Related Info — https://transplantgenomics.com/our-tests/kidney/trugraf-kidney/